CLINICAL TRIAL: NCT02253641
Title: The STRENGTH Study: Shapely Sisters Targeting Realistic Exercise and Nutrition Goals Through Healthy Habits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Academy of Nutrition and Dietetics (Other)
Responsible Party: Principal Investigator, Danielle Braxton, MPH, RD, Graduate Research Assistant, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-2107
Record Dates: First submitted 2014-09-25; First posted 2014-10-01 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Obesity
Keywords: African American, Women; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Weight Loss Intervention (Active Comparator): Participants will take part in a 14 session weight loss/healthy lifestyle intervention. Sessions will be 2 hours in length and will occur weekly for month 1 then bi-weekly for months 2 - 6. The core lifestyle curriculum content for both groups will come from the previously IRB-approved Weight Wise intervention developed by Samuel-Hodge et al. (Samuel-Hodge, Carmen D., et al. "Randomized Trial of a Behavioral Weight Loss Intervention for Low?income Women: The Weight Wise Program." Obesity 17.10 (2009): 1891-1899). The only modifications to the content (other than some general formatting) will be the combining of sessions 3 and 4 and sessions 6 and 7. These changes will allow us to fit the original 16-session curriculum into the 14-session format of our intervention.
  Interventions: Behavioral: Standard Weight Loss Intervention
- Stress-Focused Weight Loss Intervention (Experimental): Participants will take part in a 14 session weight loss/healthy lifestyle intervention. Sessions will be 2 hours in length and will occur weekly for month 1 then bi-weekly for months 2 - 6. The core lifestyle curriculum content for both groups will come from the previously IRB-approved Weight Wise intervention developed by Samuel-Hodge et al.. The participants in this arm will receive all of the content that the comparison group receives (just moderately condensed to allow time for additional components) plus a stress-reduction intervention woven into each of the sessions. The stress-reduction content aims to reduce stress by helping participants: (1) identifying and reducing exposure (to the degree possible) of current stressors, (2) change their perceptions of current stressors and (3) use healthier stress-coping techniques (e.g. yoga, meditation, etc.)
  Interventions: Behavioral: Stress-Focused Weight Loss Intervention

INTERVENTIONS:
Behavioral: Standard Weight Loss Intervention — 14-session/6-month standard behavioral weight loss intervention
  Arms: Standard Weight Loss Intervention
Behavioral: Stress-Focused Weight Loss Intervention — 14-session/6-month tailored behavioral weight loss intervention
  Arms: Stress-Focused Weight Loss Intervention

SUMMARY:
This study evaluates the efficacy of a stress-focused tailored weight loss intervention compared to a standard weight loss intervention on weight loss in severely obese (BMI > 40.0) African American women.

DETAILED DESCRIPTION:
Stress has been identified as a major barrier to engaging in healthy lifestyle behaviors (e.g. diet and exercise) among African American women. African American women consistently lose less weight than their Caucasian counterparts in weight loss interventions. One reason for this disparity may be due to the failure of most weight loss interventions to address stress management adequately or in a culturally competent way.

The purpose of this study is to evaluate the efficacy of a stress-focused tailored weight loss intervention compared to a standard weight loss intervention on weight loss in severely obese (BMI > 40.0) African American women. The stress-focused weight loss intervention will incorporate stress management content throughout the entire intervention and will include content that is culturally tailored. The standard weight loss intervention will cover stress management techniques during one of the 14 sessions and the material will be more generic in nature (e.g. not culturally tailored).

ELIGIBILITY:
Inclusion Criteria:

* African American (self-identified)
* Female
* BMI > 40 kg/m2
* Access to internet connection and phone for personal use

Exclusion Criteria:

* Unable to walk without the use of an assistance device
* Failure to pass the Physical Activity Readiness Questionnaire (PAR-Q) or unable to attain medical clearance from their doctor
* Substance abuse within past two years
* Schizophrenia
* Currently pregnant, pregnant within the past 6 months or plans to become pregnant in the next 6 months
* History of malignancy other than non-melanoma skin cancer, that has not been in remission or cured surgically for > 5 years
* Participation in a weight loss program in the past 12 months
* > 5% loss of body weight within the past 6 months
* Bariatric surgery recipient
* Heart attack in the past 6 months
* Stroke within the past 6 months

NOTE: Participants who "fail" the PAR-Q will be required to obtain medical clearance from their medical provider

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Weight | Change from Baseline to 6 Months
  collect weight in pounds

SECONDARY OUTCOMES:
Physical Activity | Change from Baseline to 6 Months
  participants will wear accelerometer for 1 week at each time point
Psychosocial & Behavioral Measures | Change from Baseline to 6 Months
  Participants will complete a survey that will assess varying psychosocial and behavioral measures including: (1) diet and exercise habits, (2) stress levels, (3) moods and (4) attitudes and beliefs regarding female stereotypes.
Walkability | Change from Baseline to 6 Months
  Stand Up and Go Test
Aerobic Fitness | Change from Baseline to 6 Months
  6 Minute Walk Test

CONTACTS AND LOCATIONS:
Locations (1):
- UNC Center for Health Promotion and Disease Prevention, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Fitzgerald KR. Review of article: Prevalence of obesity and trends in the distribution of body mass index among US adults, 1999-2010 by Katherine M. Flegal, PhD; Margaret D. Carroll, MSPH; Brian K. Kit, MD; Cynthia L. Ogden, PhD (JAMA 2012;307:491-7). J Vasc Nurs. 2013 Sep;31(3):131-2. doi: 10.1016/j.jvn.2013.06.004. No abstract available. PMID 23953862
- [Background] Goodpaster BH, Delany JP, Otto AD, Kuller L, Vockley J, South-Paul JE, Thomas SB, Brown J, McTigue K, Hames KC, Lang W, Jakicic JM. Effects of diet and physical activity interventions on weight loss and cardiometabolic risk factors in severely obese adults: a randomized trial. JAMA. 2010 Oct 27;304(16):1795-802. doi: 10.1001/jama.2010.1505. Epub 2010 Oct 9. PMID 20935337
- [Background] Ryan DH, Johnson WD, Myers VH, Prather TL, McGlone MM, Rood J, Brantley PJ, Bray GA, Gupta AK, Broussard AP, Barootes BG, Elkins BL, Gaudin DE, Savory RL, Brock RD, Datz G, Pothakamuri SR, McKnight GT, Stenlof K, Sjostrom LV. Nonsurgical weight loss for extreme obesity in primary care settings: results of the Louisiana Obese Subjects Study. Arch Intern Med. 2010 Jan 25;170(2):146-54. doi: 10.1001/archinternmed.2009.508. PMID 20101009
- [Background] West DS, Elaine Prewitt T, Bursac Z, Felix HC. Weight loss of black, white, and Hispanic men and women in the Diabetes Prevention Program. Obesity (Silver Spring). 2008 Jun;16(6):1413-20. doi: 10.1038/oby.2008.224. Epub 2008 Apr 10. PMID 18421273
- [Background] Cox TL, Krukowski R, Love SJ, Eddings K, DiCarlo M, Chang JY, Prewitt TE, West DS. Stress management-augmented behavioral weight loss intervention for African American women: a pilot, randomized controlled trial. Health Educ Behav. 2013 Feb;40(1):78-87. doi: 10.1177/1090198112439411. Epub 2012 Apr 13. PMID 22505570
- [Background] Samuel-Hodge CD, Headen SW, Skelly AH, Ingram AF, Keyserling TC, Jackson EJ, Ammerman AS, Elasy TA. Influences on day-to-day self-management of type 2 diabetes among African-American women: spirituality, the multi-caregiver role, and other social context factors. Diabetes Care. 2000 Jul;23(7):928-33. doi: 10.2337/diacare.23.7.928. PMID 10895842
- [Background] Fitzgibbon ML, Tussing-Humphreys LM, Porter JS, Martin IK, Odoms-Young A, Sharp LK. Weight loss and African-American women: a systematic review of the behavioural weight loss intervention literature. Obes Rev. 2012 Mar;13(3):193-213. doi: 10.1111/j.1467-789X.2011.00945.x. Epub 2011 Nov 10. PMID 22074195